CLINICAL TRIAL: NCT02752412
Title: A Randomized, Active-controlled, Open Label, 2-treatment Arm, and Multicenter Study Comparing the Efficacy and Safety of the Insulin Glargine/Lixisenatide Combination to Insulin Glargine With Metformin in Japanese Patients With Type 2 Diabetes Mellitus Inadequately Controlled on Basal Insulin and Oral Antidiabetic Drugs
Brief Title: Efficacy and Safety of LixiLan Versus Insulin Glargine Alone Both With Metformin in Japanese With Type 2 Diabetes Mellitus Inadequately Controlled on Basal Insulin and Oral Antidiabetic Drugs
Acronym: LIXILAN JP-L
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC14113; U1111-1176-8378 (Other: UTN)
Record Dates: First submitted 2016-04-20; First posted 2016-04-27 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2018-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; lixisenatide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LixiLan (Experimental): LixiLan (insulin glargine/lixisenatide fixed ratio combination) is injected subcutaneously (under the skin) once daily. Dose is individually adjusted.
  Metformin will be continued.
  Interventions: Drug: Insulin glargine/Lixisenatide (HOE901/AVE0010); Drug: Metformin
- insulin glargine (Active Comparator): Insulin glargine U100 (Lantus) will be injected subcutaneously (under skin) once daily. Dose will be individually adjusted.
  Metformin will be continued.
  Interventions: Drug: Insulin glargine U100 (HOE901); Drug: Metformin

INTERVENTIONS:
Drug: Insulin glargine/Lixisenatide (HOE901/AVE0010) — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: LixiLan
  Arms: LixiLan
Drug: Insulin glargine U100 (HOE901) — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: Lantus
  Arms: insulin glargine
Drug: Metformin — Pharmaceutical form: tablet
  Route of administration: oral

SUMMARY:
Primary Objective:

To compare LixiLan to insulin glargine in glycated hemoglobin (HbA1c) change from baseline to week 26 in patients with type 2 diabetes mellitus.

Secondary Objective:

To compare overall efficacy and safety of LixiLan to insulin glargine over 26 weeks in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
The maximum study duration per patient will be approximately 41 weeks: an up to 14-week screening period (consisting of an up to 2-week screening phase and a 12-week run-in phase), a 26-week randomized treatment period, and a 3-day post-treatment safety follow-up period.

ELIGIBILITY:
Inclusion criteria :

* Patient with type 2 diabetes mellitus (T2DM) diagnosed for at least 1 year before the screening visit (V1).
* Patient treated with a stable, once a day basal insulin regimen (ie, type of insulin and time/frequency of the injection), for at least 3 months before the screening visit.
* The total daily basal insulin dose should be stable (± 20%) and <15 U/day for at least 1 month before the screening visit.
* Patient receiving 1 or 2 oral anti-diabetic drugs (OADs): the OAD dose(s) must be stable during the 3 months before the screening visit. The OADs can be 1 to 2 out of:
* Metformin;
* Sulfonylurea (SU);
* Glinide;
* Dipeptidyl-peptidase-4 (DPP-4) inhibitor;
* Sodium glucose co-transporter 2 (SGLT2) inhibitor;
* Alpha glucosidase inhibitor (alpha-GI).
* Signed written informed consent.

Exclusion criteria:

* Age <20 years at screening visit.
* HbA1c at screening visit <7.5% or >9.5%.
* Fasting plasma glucose (FPG) >180 mg/dL (10.0 mmol/L) at screening visit.
* Pregnancy or lactation, women of childbearing potential with no effective contraceptive method.
* Use of oral or injectable glucose-lowering agents other than those stated in the inclusion criteria in the 3 months before screening visit.
* Previous use of insulin regimen other than basal insulin, eg, prandial or pre-mixed insulin.

Note: Short-term treatment (≤10 days) due to intercurrent illness including gestational diabetes is allowed at the discretion of the Investigator.

* Use of thiazolidinedione (TZD) within 6 months prior to screening visit.
* History of discontinuation of a previous treatment with a glucagon-like peptide-1(GLP-1) receptor agonist due to safety/ tolerability issues or lack of efficacy.
* Laboratory findings at the screening visit; including:
* Amylase and/or lipase >3 times the upper limit of the normal (ULN) laboratory range;
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 ULN;
* Calcitonin ≥20 pg/mL (5.9 pmol/L);
* Positive serum pregnancy test.
* Any contraindication to metformin use according to local labeling.
* History of hypersensitivity to any GLP-1 receptor agonist or to metacresol.
* Contraindication to use of insulin glargine or lixisenatide according to local labeling. History of hypersensitivity to insulin glargine or to any of the excipients.
* Personal or immediate family history of medullary thyroid cancer (MTC) or genetic condition that predisposes to MTC (eg, multiple endocrine neoplasia syndromes).
* History of pancreatitis (unless pancreatitis was related to gallstones and cholecystectomy has now been performed), pancreatitis during previous treatment with incretin therapies, chronic pancreatitis, pancreatectomy, stomach/gastric surgery.
* Exclusion criteria for randomization at the end of the run-in phase:
* HbA1c <7.5% or >9.5% at visit 6 (Week -1).
* Mean fasting self monitored plasma glucose (SMPG) >160 mg/dL (8.9 mmol/L), calculated from all available (minimum of 4 self-measurements) values during the 7 days prior to randomization.

Note:fasting SMPG on the day of randomization can be included if assessed before randomization.

* Average insulin glargine daily dose ≥15 U/day or <5U/day calculated for the last 3 days before Visit 7.
* Metformin total daily dose <750 mg/day.
* Amylase and/or lipase >3 ULN at Visit 6 (Week -1).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2016-05-17 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | Baseline, 26 weeks

SECONDARY OUTCOMES:
Percentage of patients reaching HbA1c <7% or ≤6.5% | 26 weeks
Change from baseline in 2-hour postprandial plasma glucose (PPG) during standardized meal test | Baseline, 26 weeks
Change from baseline in blood glucose excursion during standardized meal test | Baseline, 26 weeks
Change from baseline in 7-point self-monitoring plasma glucose (SMPG) profiles (each time point and average daily value) | Baseline, 26 weeks
Change from baseline in body weight | Baseline, 26 weeks
Change from baseline in FPG | Baseline, 26 weeks
Change from baseline in daily dose of insulin glargine | Baseline, 26 weeks
Percentage of patients reaching HbA1c <7% with no body weight gain | 26 weeks
Percentage of patients reaching HbA1c <7% with no body weight gain and with no documented (PG ≤70 mg/dL [3.9 mmol/L]) symptomatic hypoglycemia | 26 weeks
Percentage of patients reaching HbA1c <7% with no documented (PG ≤70 mg/dL [3.9 mmol/L]) symptomatic hypoglycemia | 26 weeks
Percentage of patients requiring a rescue therapy | 26 weeks
Number of hypoglycemic events | 26 weeks
Number of adverse events | 26 weeks
Measurement of anti-lixisenatide antibodies from baseline | Baseline, 26 weeks
Measurement of anti-insulin antibodies from baseline | Baseline, 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (122):
- Japan (122):
  - Investigational Site Number 392002, Adachi-Ku
  - Investigational Site Number 392132, Annaka-Shi
  - Investigational Site Number 392009, Arakawa-Ku
  - Investigational Site Number 392152, Asahikawa-Shi
  - Investigational Site Number 392025, Atsugi-Shi
  - Investigational Site Number 392024, Chiba
  - Investigational Site Number 392151, Chiba
  - Investigational Site Number 392011, Chigasaki-Shi
  - Investigational Site Number 392013, Chiyoda-Ku
  - Investigational Site Number 392052, Chiyoda-Ku
  - Investigational Site Number 392003, Chūōku
  - Investigational Site Number 392017, Chūōku
  - Investigational Site Number 392055, Chūōku
  - Investigational Site Number 392008, Fujimi-Shi
  - Investigational Site Number 392143, Fujisawa-Shi
  - Investigational Site Number 392094, Fukuoka
  - Investigational Site Number 392147, Fukuoka
  - Investigational Site Number 392100, Gifu
  - Investigational Site Number 392059, Hachioji-Shi
  - Investigational Site Number 392048, Hamamatsu
  - Investigational Site Number 392102, Hamamatsu
  - Investigational Site Number 392123, Higashiosaka-Shi
  - Investigational Site Number 392135, Higashiosaka-Shi
  - Investigational Site Number 392079, Hiki-Gun
  - Investigational Site Number 392141, Himeji-Shi
  - Investigational Site Number 392057, Iruma-Shi
  - Investigational Site Number 392022, Ise-Shi
  - Investigational Site Number 392020, Izumisano
  - Investigational Site Number 392036, Kamakura-Shi
  - Investigational Site Number 392136, Kamogawa-Shi
  - Investigational Site Number 392066, Kashiwa-Shi
  - Investigational Site Number 392045, Kashiwara-Shi
  - Investigational Site Number 392006, Kasugai-Shi
  - Investigational Site Number 392149, Kasugai-Shi
  - Investigational Site Number 392053, Kawagoe-Shi
  - Investigational Site Number 392065, Kawagoe-Shi
  - Investigational Site Number 392007, Kawaguchi-Shi
  - Investigational Site Number 392062, Kawaguchi-Shi
  - Investigational Site Number 392090, Kawaguchi-Shi
  - Investigational Site Number 392077, Kawasaki-Shi
  - Investigational Site Number 392082, Kawasaki-Shi
  - Investigational Site Number 392142, Kawasaki-Shi
  - Investigational Site Number 392010, Kisarazu-Shi
  - Investigational Site Number 392016, Kisarazu-Shi
  - Investigational Site Number 392031, Kitakyushu-Shi
  - Investigational Site Number 392068, Kitakyushu-Shi
  - Investigational Site Number 392041, Kitakyusyu-Shi
  - Investigational Site Number 392086, Kobe
  - Investigational Site Number 392044, Koga-Shi
  - Investigational Site Number 392001, Koriyama-Shi
  - Investigational Site Number 392028, Kumamoto
  - Investigational Site Number 392092, Kumamoto
  - Investigational Site Number 392108, Kumamoto
  - Investigational Site Number 392116, Kumamoto
  - Investigational Site Number 392099, Kushiro
  - Investigational Site Number 392049, Kyoto
  - Investigational Site Number 392107, Kyoto
  - Investigational Site Number 392088, Maebashi
  - Investigational Site Number 392158, Maebashi
  - Investigational Site Number 392121, Matsuyama
  - Investigational Site Number 392122, Minatoku
  - Investigational Site Number 392076, Misato-Shi
  - Investigational Site Number 392014, Mitaka-Shi
  - Investigational Site Number 392042, Mito
  - Investigational Site Number 392043, Mito
  - Investigational Site Number 392078, Mito
  - Investigational Site Number 392046, Miyazaki
  - Investigational Site Number 392026, Nagoya
  - Investigational Site Number 392101, Nagoya
  - Investigational Site Number 392128, Nagoya
  - Investigational Site Number 392131, Nagoya
  - Investigational Site Number 392134, Nagoya
  - Investigational Site Number 392137, Nagoya
  - Investigational Site Number 392140, Nagoya
  - Investigational Site Number 392154, Naka
  - Investigational Site Number 392050, Niihama-Shi
  - Investigational Site Number 392159, Obihiro-Shi
  - Investigational Site Number 392145, Ogaki-Shi
  - Investigational Site Number 392005, Okawa-Shi
  - Investigational Site Number 392071, Okayama
  - Investigational Site Number 392080, Okayama
  - Investigational Site Number 392095, Onga-Gun
  - Investigational Site Number 392105, Osaka
  - Investigational Site Number 392117, Osaka
  - Investigational Site Number 392144, Osaka
  - Investigational Site Number 392125, Osaki-Shi
  - Investigational Site Number 392157, Ota-Shi
  - Investigational Site Number 392040, Oyama-Shi
  - Investigational Site Number 392153, Ōita
  - Investigational Site Number 392120, Ōta-ku
  - Investigational Site Number 392038, Sagamihara-Shi
  - Investigational Site Number 392069, Saijo-Shi
  - Investigational Site Number 392030, Saitama-Shi
  - Investigational Site Number 392058, Saitama-Shi
  - Investigational Site Number 392074, Sanda-Shi
  - Investigational Site Number 392047, Sapporo
  - Investigational Site Number 392106, Sapporo
  - Investigational Site Number 392097, Sasebo-Shi
  - Investigational Site Number 392015, Satsumasendai-Shi
  - Investigational Site Number 392004, Sendai
  - Investigational Site Number 392034, Shimotsuke-Shi
  - Investigational Site Number 392110, Shinagawa-Ku
  - Investigational Site Number 392021, Shinjuku-Ku
  - Investigational Site Number 392098, Shinjuku-Ku
  - Investigational Site Number 392104, Shiogama-Shi
  - Investigational Site Number 392037, Shizuoka
  - Investigational Site Number 392081, Shizuoka
  - Investigational Site Number 392019, Shobara-Shi
  - Investigational Site Number 392018, Shunan-Shi
  - Investigational Site Number 392027, Suita-Shi
  - Investigational Site Number 392056, Taito-Ku
  - Investigational Site Number 392051, Takatsuki-Shi
  - Investigational Site Number 392156, Takatsuki-Shi
  - Investigational Site Number 392061, Tokorozawa-Shi
  - Investigational Site Number 392111, Tomakomai-Shi
  - Investigational Site Number 392073, Tsu
  - Investigational Site Number 392063, Ube-Shi
  - Investigational Site Number 392124, Ushiku-Shi
  - Investigational Site Number 392067, Yatsushiro-Shi
  - Investigational Site Number 392085, Yokohama
  - Investigational Site Number 392126, Yokohama
  - Investigational Site Number 392035, Zentsuji-Shi

REFERENCES:
- [Result] Kaneto H, Takami A, Spranger R, Amano A, Watanabe D, Niemoeller E. Efficacy and safety of insulin glargine/lixisenatide fixed-ratio combination (iGlarLixi) in Japanese patients with type 2 diabetes mellitus inadequately controlled on basal insulin and oral antidiabetic drugs: The LixiLan JP-L randomized clinical trial. Diabetes Obes Metab. 2020 Sep;22 Suppl 4:3-13. doi: 10.1111/dom.14005. PMID 32072742